CLINICAL TRIAL: NCT02781025
Title: Culture of Circulating Tumor Cells Isolated From Cancer Patients With Metastatic Disease
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1604
Record Dates: First submitted 2016-05-10; First posted 2016-05-24 (Estimated); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Circulating Tumor Cells
MeSH Terms: conditions — Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Oligometastatic Disease: Patients with oligometastatic cancer, defined as biopsy proven disease involving at least one organ other than the primary tumor organ. Regional lymph node metastases are not considered metastatic.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — A blood sample of 10mL- 25mL will be collected before the start of radiation treatment.

SUMMARY:
The purpose of this study is to investigate the feasibility of using novel decellularized tissue matrices to isolate and culture circulating tumor cells (CTCs) collected from patients with metastatic solid tumor malignancies.

DETAILED DESCRIPTION:
There are currently very few practical or reproducible model systems which recapitulate the metastatic process well. CTCs are important for the development of metastases and there is interest in isolating and culturing them ex vivo to better characterize their biology, metastatic potential, and response to different therapies. The investigators have previously demonstrated efficient capture and enumeration of CTCs in 4 unique patient cohorts (metastatic prostate and locally advanced rectal, cervical and head and neck cancers) in the investigators prospective clinical study, LCCC 1408 (Investigation of Circulating Tumor Cells from Cancer Patients Undergoing Radiation Therapy). However, CTCs are difficult to culture with conventional methods. The investigators propose to culture CTCs using novel decellularized tissue matrices. Blood will be collected from cancer patients with metastatic solid tissue tumors prior to starting definitive or palliative radiotherapy. The investigators will then isolate CTCs and attempt to grow them on various decellularized matrices. If this study is successful and feasibility is demonstrated, important pilot information will also be gathered which will then be used in power and sample size considerations for future CTCs studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any metastatic solid tumor malignancy. Metastatic is defined as biopsy proven disease involving at least one organ other than the primary tumor organ. Regional lymph node metastases are not considered metastatic. Patients with newly diagnosed metastatic disease who have not had systemic therapy in at least six months or are progressing on systemic therapy will be eligible for enrollment.
* Scheduled to initiate radiation for management of their disease, and schedule accommodates blood sample collection prior to radiation
* Male and female of ≥18 years of age
* Male and female patients capable of reproduction must agree to use medically acceptable methods of contraception, such as an intra-uterine device, diaphragm, with spermicide, condom with spermicide or abstinence, during radiation therapy. Inclusion of females of childbearing potential requires a negative pregnancy test within 14 days prior to study initiation (part of standard of care in radiation oncology).
* Written informed consent obtained and signed
* Able to have blood collection without excessive difficulty

Exclusion Criteria:

* Patient unwilling or unable to complete informed consent
* Physical or psychological inability to complete sample collection for any reason including but not limited to: inability to tolerate any study procedures, any physical limitation that would undermine the safety of the subject in the study, or any psychiatric or neurological condition that inhibits full comprehension of study requirements and inability to complete informed consent, as determined by treating physician
* Currently pregnant or lactating women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing radiation treatments at Lineberger Comprehensive Cancer Center at UNC Hosptials for treatments of oligometastatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2016-04; Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
The proportion of successful CTC culture growths. | through study completion, an average of 6 months
  The proportion of successful CTC culture growths will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wang, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org/